CLINICAL TRIAL: NCT03826043
Title: "Prospective Study Evaluating the Impact and Treatment of Thrombo-embolic Events in Patients With Cancer"
Brief Title: THrombo-Embolic Event in Onco-hematology
Acronym: THEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/23; 2018-A01120-55 (Other: ANSM ID RCB)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms; Thrombosis; Coagulation Disorder
Keywords: Neoplasms, Thrombosis, hypocoagulability
MeSH Terms: conditions — Neoplasms; Thrombosis; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Hospitalized patient
  Interventions: Diagnostic Test: Blood sample analysis

INTERVENTIONS:
Diagnostic Test: Blood sample analysis — Thrombophilia, blood count and coagulation count

SUMMARY:
The overall incidence of deep vein thrombosis (DVT) and pulmonary embolism (PE) is 1 per 200 cancer patients, about 5 times higher than in the general population.

These events are of crucial importance, since nearly 10% of cancer patients died from thromboembolic events (EVT), making them the second leading cause of death in this population.

In hospitalized patients, the rate seems to have increase between 1979 and 1990 from 0.6% - 2% before 1990 to 4% since 1990.

Thrombotic risk in cancer patients is known and identified. Thrombotic complications affect the survival and quality of life of cancer patients.

Chemotherapy is a regular generator of cytopenia, the most prominent of which is thrombocytopenia. In addition, a prospective study of 107 cancer patients in our institution shows that almost 40% of patients over 65 years of age take anticoagulant or antiplatelet therapy.

In this specific population (i.e., with cancer and hypocoagulability), the occurrence of thrombosis poses particular problems. The prevalence and incidence of venous thrombosis in this situation is unknown and the behavior to be poorly specified.

Based on these considerations, The investigator propose a two-year prospective cohort study to explore the biological parameters of hypocoagulability and to assess the incidence and prevalence of DVT in thrombocytopenic patients on vitamin K antagonists. (AVK), anti-platelet aggregation (AGP) and / or direct oral anticoagulant (AOD).

In this study, the investigator means by hypocoagulability any situation modifying the normal coagulation system.

DETAILED DESCRIPTION:
The overall incidence of deep vein thrombosis (DVT) and pulmonary embolism (PE) is 1 per 200 cancer patients, about 5 times higher than in the general population.

These events are of crucial importance, since nearly 10% of cancer patients died from thromboembolic events (EVT), making them the second leading cause of death in this population.

In hospitalized patients, the rate seems to have increase between 1979 and 1990 from 0.6% - 2% before 1990 to 4% since 1990.

Some studies report an increase in the hospitalization cost of 38%, correlated in part with the increase in hospitalization duration related to venous thromboembolism.

Thrombotic risk in cancer patients is known and identified. Thrombotic complications affect the survival and quality of life of cancer patients. Scores were established and validated to establish this risk and to propose prophylaxis in these patients. Guidelines exist for prophylaxis and for the treatment of these patients.

Chemotherapy is a regular generator of cytopenia, the most prominent of which is thrombocytopenia. In addition, a prospective study of 107 cancer patients in our institution shows that almost 40% of patients over 65 years of age take anticoagulant or antiplatelet therapy.

In this specific population (i.e., with cancer and hypocoagulability), the occurrence of thrombosis poses particular problems. The prevalence and incidence of venous thrombosis in this situation is unknown and the behavior to be poorly specified.

Based on these considerations, The investigator propose a two-year prospective cohort study to explore the biological parameters of hypocoagulability and to assess the incidence and prevalence of DVT in thrombocytopenic patients on vitamin K antagonists. (AVK), anti-platelet aggregation (AGP) and / or direct oral anticoagulant (AOD).

In this study, the investigator means by hypocoagulability any situation modifying the normal coagulation system, that is to say:

* The presence of any anti-coagulant or antiplatelet treatment,
* Or abnormalities of primary or secondary hemostasis causing coagulation disorders.

Some studies report an increase in the hospitalization cost of 38%, correlated in part with the increase in hospitalization duration related to venous thromboembolism.

Thrombotic risk in cancer patients is known and identified. Thrombotic complications affect the survival and quality of life of cancer patients. Scores were established and validated to establish this risk and to propose prophylaxis in these patients. Guidelines exist for prophylaxis and for the treatment of these patients.

Chemotherapy is a regular generator of cytopenia, the most prominent of which is thrombocytopenia. In addition, a prospective study of 107 cancer patients in our institution shows that almost 40% of patients over 65 years of age take anticoagulant or antiplatelet therapy.

In this specific population (i.e., with cancer and hypocoagulability), the occurrence of thrombosis poses particular problems. The prevalence and incidence of venous thrombosis in this situation is unknown and the behavior to be poorly specified.

Based on these considerations, The investigator propose a two-year prospective cohort study to explore the biological parameters of hypocoagulability and to assess the incidence and prevalence of DVT in thrombocytopenic patients on vitamin K antagonists (AVK), anti platelet aggregation (AGP) and / or direct oral anticoagulant (AOD).

In this study the investigator mean by hypocoagulability any situation modifying the normal coagulation system, that is to say:

* the presence of any anti-coagulant or antiplatelet treatment,
* or abnormalities of primary or secondary hemostasis causing coagulation disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Patient followed for CAL cancer and admitted to the LTC in the Medicine Department.
2. Age> to 18 years.
3. Patient having read the information note and signed the informed consent (including specific consent for genotyping of clotting factors).
4. Patient receiving social insurance.
5. Weight> 50kg
6. Hemoglobin level> 7.0 g / dl

Exclusion Criteria:

1. Patient not benefiting as part of his treatment from hospitalization, but admitted on an ambulatory basis.
2. Patient whose age is less than 18 years.
3. Patient already included in the study.
4. Patient considered a vulnerable person; Vulnerable people are defined in Article L1121-5 to -8:

   * Pregnant women, parturients and breastfeeding mothers
   * Persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent under Articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of Article L. 1121-8
   * and persons admitted to a health or social institution for purposes other than research
   * adults who are legally protected or unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of thrombosis rate in patients hospitalized for cancer | 12 months
  Incidence rate of first occurrence of thromboembolic event in cancer patients, and hospitalized

SECONDARY OUTCOMES:
Comparison of the values of the biological parameters of thrombophilia assessment, blood count and coagulation, at the time of the occurrence of thrombosis, between patients in a situation of hypocoagulability and patients with no hypocoagulability. | 12 months
  These patients in these two situations, will be identified, during the onset of thrombosis, the results of the parameters of their blood count and their intake of antiaggregant or anticoagulant treatment.
  • Comparison between the hypocoagulable patient group and the non-hypocoagulable patient group of the biological parameters of the thrombophilia balance, blood counts and coagulation counts in patients with cancer at the time of the occurrence of thrombosis
  o The state of hypocoagulability is defined by: thrombocytopenia <100000 / mm3, abnormality of one or more coagulation factors, platelet antiaggregant treatment, anticoagulant treatment of all kinds.
Determination of thrombosis rate with new oral anticoagulants. | 12 months
  Incidence rate of first occurrence of thromboembolic events in patients with cancer, and treatment with new oral anticoagulants
Comparison of 12-month survival of patients with or without hypocoagulability, with thrombosis. | 12 months
  Survival at 12 months. 12-month survival is defined as the delay between the date of inclusion and the date of death from all causes. Patients lost to follow-up will be censored on the date of the latest news. Patients will be followed for 12 months after inclusion in the study.
• Determination of death rate due to thrombosis. | 12 months
  Death rate due to thrombosis is the number of deaths whose cause is thrombosis.
Determination of the rate of hemorrhagic complications in this population. | 12 months
  Rate of haemorrhagic complications defined by the number of haemorrhagic events, whatever the degree of severity, of biological or medicinal origin.
  o A haemorrhagic event is defined as the occurrence of bleeding by rupture of a blood vessel or effusion out of a blood vessel. Bleeding may be internal or external, see the examples provided below: Internal haemorrhage: cerebral hematoma, subdural hematoma; intramuscular hematoma
  - Externalized hemorrhage: epistaxis, gingivorrhagia, externalized digestive bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No